CLINICAL TRIAL: NCT03675048
Title: Single-center, Prospective, Randomized, Double-blind, Placebo-controlled Clinical Trial on Estimating the Effect of Probiotic Strain Lactobacillus Reuteri DSM 17938 on Gut Microbiota Modulation in Infants Born by Caesarean Section
Brief Title: Lactobacillus Reuteri DSM 17938 in Gut Microbiota Development in Infant Born by Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSUB0142
Record Dates: First submitted 2018-09-14; First posted 2018-09-18 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Dysbiosis; Prophylaxis
Keywords: Gut Microbiota; Cesarean Section; Dysbiosis
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): The intervention group will receive 5 drops (10^8 cfu Lactobacillus reuteri DSM 17938) twice daily during feeding for 4 weeks.
  Interventions: Dietary Supplement: BioGaia Protectis drops
- Placebo group (Placebo Comparator): The placebo group will receive 5 drops twice daily during feeding for 4 weeks. Placebo composition will be identical to that of the study drug but will not contain L. reuteri.
  Interventions: Dietary Supplement: Placebo
- Control group (No Intervention): The infants from the control group will comply with the same requirements and will undergo the same procedures as participants from the main group except for randomization and treatment.

INTERVENTIONS:
Dietary Supplement: BioGaia Protectis drops — food supplement containing the patented lactic acid bacterium Lactobacillus reuteri Protectis®/™ (L. reuteri DSM 17938).
  Other Names: BioGaia® Probiotic. Drops for baby
  Arms: Intervention group
Dietary Supplement: Placebo — Contains same excipients as study drug, without the active ingredient L. Reuteri.
  Arms: Placebo group

SUMMARY:
The aim of this study is to assess influence of probiotic Lactobacillus reuteri DSM 17938 on formation of gut microbiota in infant born by Caesarean section. It is anticipated that daily using of probiotic Lactobacillus reuteri DSM 17938 can prevent development of early dysbiosis of gut microbiota induced by Caesarean section.

DETAILED DESCRIPTION:
This is a single-center prospective randomized double-blind placebo-controlled clinical study. The planned duration of the study for each included infant will be 16 weeks, 4 weeks of study drug intake and 12 weeks of follow-up. 140 healthy infants born by Caesarean section will be included in the general group of the study, and 60 healthy infants born by natural vaginal delivery will be included in the control group. For infants included in the control group, all the same protocol requirements and procedures will be applied as for infants in the general group, except for randomization and the study product / placebo intake. Infants included in the general study group will be randomly assigned into the study product / placebo subgroups in 1: 1 ratio. During the study the gut microbiota will be analyzed. Feces samples should be collected no later than 72 hours after birth, and also on 14th day of life ± 3 days, 30th day of life ± 3 days and 112th day of life ± 3 days. Short-chain fatty acids (SCFA) will be analyzed in feces samples.

ELIGIBILITY:
Inclusion Criteria:

* gestational age more than 37 weeks and less than 41 weeks
* age of enrolment is not more than 48 hours
* birth weight is corresponded to gestational age
* Apgar score ≥8 at 5 minutes
* Absence of congenital anomaly and/or clinical or physical abnormalities identified during clinical examination
* Primarily breastfeeding during the first days of life (more than 50%)
* Parent(s) are willing to comply with the exclusive breastfeeding regime during study period
* Parent(s) are willing to follow dietary recommendations during study period
* Parent(s) are willing to fill in the Diary every day
* Availability of the parent(s) and the infant during study period
* Written informed consent of the parent(s)

Exclusion Criteria:

* Chronic diseases or serious health problems of mother or child
* Gastrointestinal tract diseases of mother or child
* Delay in development
* Congenital abnormalities
* Intake of antibiotics by mother orally and / or vaginally during the last trimester of pregnancy
* Intake of probiotics by mother during the last trimester of pregnancy
* Using of general anesthesia during Caesarean section
* Emergency Caesarean section

Ages: 0 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Composition of gut microbiota in infants born by Caesarean section | 14 days
  Composition of gut microbiota in infants born by Caesarean section in group received L. reuteri DSM 17938 versus placebo group at 14+/-3 day after delivery.

SECONDARY OUTCOMES:
Composition of gut microbiota in infants born by vaginal delivery | 14 days
  Composition of gut microbiota in infants born by vaginal delivery in comparison with infants born by Caesarean section and received L. reuteri DSM 17938 at 14+/-3 day after delivery.
Composition of gut microbiota in infants born by vaginal delivery | 30 days
  Composition of gut microbiota in infants born by vaginal delivery in comparison with infants born by Caesarean section and received L. reuteri DSM 17938 at 30+/-3 day after delivery.
Composition of gut microbiota in infants born by Caesarean section | 30 days
  Composition of gut microbiota in infants born by Caesarean section in group received L. reuteri DSM 17938 versus placebo group at 30+/-3 day after delivery.
Composition of gut microbiota in infants born by Caesarean section | 112 days (16 weeks)
  Composition of gut microbiota in infants born by Caesarean section in group received L. reuteri DSM 17938 versus placebo group at 112+/-3 day (16 weeks) after delivery.
Composition of gut microbiota in infants born by vaginal delivery | 112 days (16 weeks)
  Composition of gut microbiota in infants born by vaginal delivery in comparison with infants born by Caesarean section and received L. reuteri DSM 17938 at 112+/-3 day (16 weeks) after delivery.
Composition of short-chain fatty acids (SCFA) in infants born by vaginal delivery | 14 days
  Composition of short-chain fatty acids in infants born by vaginal delivery in comparison with infants born by Caesarean section and received L. reuteri DSM 17938 at 14+/-3 day after delivery.
Composition of short-chain fatty acids (SCFAs) in infants born by Caesarean section | 14 days
  Composition of short-chain fatty acids in infants born by Caesarean section in group received L. reuteri DSM 17938 versus placebo group at 14+/-3 day after delivery.
Adverse events assessment | 112 days (16 weeks)
  Incidence of adverse events observed during usage of L. reuteri DSM 17938 in drop form.

CONTACTS AND LOCATIONS:
Locations (1):
- State Autonomous Healthcare Institution of the Moscow Region "Central clinical hospital of Khimki", Khimki, Moscow Oblast, Russia